CLINICAL TRIAL: NCT07102342
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Feasibility, and Preliminary Efficacy of NouvNeu001 in Patients With Advanced Parkinson's Disease.
Brief Title: This Clinical Trial is Designed to Evaluate the Safety, Tolerability, Feasibility and Preliminary Efficacy of NouvNeu001 (Human Dopaminergic Progenitor Cells Injection) in Patients With Parkinson's Disease.
Acronym: NouvNeu001-01
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: iRegene Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NouvNeu001-01
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: NouvNeu001; Human Dopaminergic Progenitor Cells Injection; phase 1 study; Dopaminergic Progenitor Cells
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NouvNeu001 (Experimental): Single injection of Human Dopaminergic Progenitor Cells into the bilateral putamen/striatum regions of the brain.
  Interventions: Biological: Human Dopaminergic Progenitor Cells

INTERVENTIONS:
Biological: Human Dopaminergic Progenitor Cells — Single injection of Human Dopaminergic Progenitor Cells into the biliteral putamen/striatum regions of the brain
  Other Names: NouvNeu001

SUMMARY:
This is a phase 1 clinical study to evaluate the safety, tolerability, feasibility, and preliminary efficacy of NouvNeu001 in patients with advanced Parkinson's Disease.

DETAILED DESCRIPTION:
This is a multi-center, single arm, and open label trial. The NouvNeu001 will be transplanted into the bilateral putamen/striatum using stereotactic neurosurgery. Subjects will take immunosuppressants to prevent potential immune rejection for 24 to 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

Age

• Male or female patient must be 30 to 75 years of age inclusive, at the time of signing the informed consent form (ICF).

Type of Patient and Disease Characteristics

* Diagnosis of PD between past 4 to 20 years (meet MDS 2015 clinical diagnostic criteria for PD).
* H-Y staging (Appendix III) for "OFF" episodes is 2.5-4.0.
* MDS-UPDRS-III score > 35, and positive for the Acute levodopa challenge test (ALCT) (improvement > 30% for MDS UPDRS-III staging from OFF episodes to ON episodes) over two screening period visits. Baseline scores will be computed as the means of two screening period visits.
* No significant change in UPDRS-III scores between the two visits during the screening period.
* Patients who take stable doing of dopamine drug for at least 4 weeks prior to receiving the study drug.
* No significant change in dose and dosing schedule of the prescribed medicines for PD during the screening period.
* Medically suitable for neurosurgery under general anesthesia.
* Acceptable laboratory test values during screening and prior to transplantation (Day 0):

  * Absolute neutrophil count ≥ 2.0 × 109/L
  * White blood cell count ≥ 4.0 × 109/L
  * Platelet count ≥ 100 × 109/L
  * Aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN)
  * Total bilirubin ≤ 1.5 x ULN
  * Serum creatinine ≤ 1.5 x ULN
  * eGFR ≥ 50 mL/min/1.73 m2
* Agree to postpone any additional neurosurgical procedures, including DBS, until completion of the 12-month follow-up study (unless recommended by a neurologist).
* Agree not to participate in any other therapeutic intervention study within 24 months after neurosurgery.
* Able to participate in all study visits and evaluations, including brain/spine MRI, CT and PET scan.

Weight • Body mass index (BMI) within the range of 18~32 kg/m2 (inclusive) with a minimum body weight of 45 kg at screening.

Sex and Contraceptive/Barrier Requirements

• Contraceptive use by men and women for 12 months after neurosurgery should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Informed Consent

* Able to understand the rationale of the clinical trial and sign the ICF. Other Inclusion Criteria
* Agree not to receive COVID-19 vaccine within 14 days before neurosurgery, and not to receive any other vaccine within 30 days after neurosurgery

Exclusion Criteria:

Medical Conditions

* Atypical Parkinsonism (Parkinsonism-Plus syndrome, secondary parkinsonism, familial parkinsonism) Prior/Concomitant Therapy
* Patients who have had previous pallidotomy, DBS surgery, striatal or extrapyramidal surgery, brain stereotaxy, prior surgical or radiation therapy to the brain or spinal cord, or other brain surgery; as well as other surgical procedures that, in the investigator's judgment, could interfere with participation in this study.
* Patients who have a previous head CT/MRI examination showing cerebral trauma, vascular malformation, hydrocephalus, brain tumor, etc., and patients who have brain imaging abnormalities in the striatum or other brain areas leading to a significantly increased risk for surgery.
* Patients who have had previous cellular therapy.
* Patients who have used glucocorticoids for an extended period (≥14 days) and at high doses (equivalent to prednisone ≥ 20 mg/day or other glucocorticoids at equivalent doses) within 3 months prior to signing the ICF. (excluding topical treatment)
* Patients who have used immunosuppressive drugs for an extended period (≥14 days) within 3 months prior to signing the ICF.
* Patients who have used antipsychotics, such as antidepressants, antimanic drugs, etc. within 3 months prior to signing the ICF and are deemed by the investigator to potentially impact the study assessment.
* Patients who have used botulinum toxin or other drugs for dystonia or muscle spasticity within 6 months prior to signing the ICF and are deemed by the investigator to potentially impact the study assessment.

Prior/Concurrent Clinical Study Experience

* Patients who are participating in other clinical trials, or have been enrolled in other clinical studies within 3 months prior to the screening
* Patients with poor compliance based on clinical evaluation of the investigator. Diagnostic Assessments
* Patients with a history of dementia or a severe cognitive disorder; or those with obvious dementia or congnitive impairment detected during screening; MDS-UPDRS congnitive impairment score (section 1.1) > 3 point at screening; or patinets with poor compliance, inability to accurately keep diary, and/or inability to sign ICF due to dementia.
* Severe depression as defined by HAMD ≥ 24 at screening.
* Severe anxiety as defined by HAMA ≥ 29 at screening.
* Patients with a history of psychiatric disorders that, in the investigator's opinion, make them unsuitable for participation; or patients with a history of suicidal ideation or suicide attempts within the past year or currently (including actual attempts, interrupted attempts, or failed attempts).
* Patients with abnormal coagulation (prothrombin time ≥ 1.5 ULN, activated partial thromboplastin time ≥ 1.5 ULN), or abnormal INR at screening.
* Patients cannot temporarily suspend anti-platelet agents or other anti-coagulant medications at least 5 days prior to investigational drug administration surgery.
* Patients with active disseminated intravascular coagulation and significant hemorrhagic tendency within 3 months prior to signing the ICF.
* Patients with current or history of following disease

  * severe heart failure (congestive heart failure of New York Heart Association Class II or above), unstable angina pectoris, and myocardial infarction
  * severe arrhythmia, including but not limited to second- or third-degree atrioventricular block, or prolonged QT interval.
  * Long QT Syndrome.
  * cardiovascular surgery (cardiac, vascular stent surgery, angioplasty).
  * stroke or transient ischemic attack within 3 months prior to signing the ICF, as determined by the investigator to be unsuitable to participate the study.
  * subarachnoid hemorrhage
  * primary mitochondrial disorder, multiple sclerosis, or other neurodegenerative diseases such as Alzheimer's disease
  * major vascular diseases (aortic aneurysm, aortic dissecting aneurysm, internal carotid artery stenosis), as determined by the investigator to be unsuitable to participate the study.
  * previous or current malignant tumors
  * immune disfunction, including autoimmune disease or immunocompromised state
  * traumatic brain injury with loss of consciousness and residue neurologic symptoms
  * active epilepsy or currently on anti-epileptic drugs
* Hypertensive patients with poorly controlled blood pressure (defined as blood pressure above 160/100 mmHg despite antihypertensive drugs treatment) and patients with severe postural hypotension
* Diabetic patients with poorly controlled blood glucose (glycosylated hemoglobin > 9.0%, or fasting plasma glucose (FPG) ≥ 11.1mmol/L)
* Patients with clinically significant abnormalities in kidney or liver function at screening.
* Patient with clinically significant abnormalities in immunological tests at screening
* Patients with surgical contraindications (such as those with cochlear implant, cardiac pacemaker, cardiac defibrillator, stereotactic nucleus pallidotomy; Patients who have had unilateral or bilateral intraparenchymal implantation of cellular products, or other surgical procedures within 6 months before screening which, in the opinion of the investigator, have an impact on this trial; Patients with other neurosurgical contraindications)
* Patients with other combined severe systemic diseases, such as pulmonary heart disease, moderate to severe asthma, severe chronic obstructive pulmonary disease (COPD) (FEV1% < 50%)
* Patients with serious infections, requiring antibiotic treatment within 2 weeks prior to signing the ICF
* Patients with any active infectious disease, including but not limited to positive for human immunodeficiency virus, SARS Covid-19 virus, syphilis antibody, quantitative HCV-RNA testing, quantitative HBV-DNA testing greater than normal range for test results, or untreated tuberculosis; any other active infection that, in the investigator's opinion, may affect the participant's ability to take part in the study or could impact study outcomes.

Other Exclusion Criteria

* Patients with alcohol or drug addiction
* Patients with contraindications or a history of allergy to any medicines used during the neurosurgical procedure.
* Patients with contraindication or a history of allergy to any medicines used during the study, such as immunosuppressants, levodopa, etc, or any of their components; Patients who are allergic to similar drugs or other macrolides.
* Female of childbearing potential who are not surgically sterilized/premenopausal/unwilling to use medically approved effective contraception during the study and lactating women; men who are not surgically sterilized/unwilling to use medically approved effective contraception during the study
* Patients who have received electric shock therapy within 30 days prior to the investigational drug administration surgery
* Patients who are participating in other clinical trials, or have been enrolled in other clinical studies within 3 months prior to the screening
* Patients with poor compliance based on clinical evaluation of the investigator
* Patients who are being treated with drugs such as neuroleptics, apomorphine, or levodopa/carbidopa infusion therapy
* Patients with severe dyskinesia in both "ON" and "OFF" drug states
* Patients who have received or will receive a live vaccine within 4 weeks prior to the study
* Patients with significant medical conditions, or with other conditions that, in the opinion of the investigator, are unsuitable to participate in the study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 24 weeks and 48 weeks post-transplant
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs).

SECONDARY OUTCOMES:
The Motor Function and Non-motor Function | 48 weeks and 96 weeks post-transplant
  Changes in MDS-UPDRS Part I-IV Score from baseline to 48 weeks and 96 weeks post-transplant. A higher score indicates more severe symptoms or worse health.
Continued Safety and Tolerability | 96 weeks and 15 years post-transplant
  Incidence and severity of AEs and SAEs within 96 weeks and 15 years post-transplant.

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell University Weill Medical College, New York, New York, United States